CLINICAL TRIAL: NCT02821312
Title: A Phase I, Randomised, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate Safety, Tolerability and Pharmacokinetics After Single and Multiple Oral Administration of DA-8010 in Healthy Subjects
Brief Title: A Study to Evaluate Safety, Tolerability and Pharmacokinetics of DA-8010 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA8010_OAB_I
Record Dates: First submitted 2016-06-19; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — DA-8010

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active in Group A1~A7 (Active Comparator): In each of Groups A1 to A7, 8 subjects will receive DA-8010.
  Interventions: Drug: DA-8010
- Placebo in Group A1~A7 (Placebo Comparator): In each of Groups A1 to A7, 2 subjects will receive placebo.
  Interventions: Drug: Placebo
- Active in Group B1~B4 (Active Comparator): In each of Groups B1 to B4, 8 subjects will receive DA-8010.
  Interventions: Drug: DA-8010
- Placebo in Group B1~B4 (Placebo Comparator): In each of Groups B1 to B4, 2 subjects will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DA-8010 — Part A will comprise a single-dose, sequential-group study incorporating a food effect evaluation. Total 70 subjects will be studied in 7 groups (Groups A1 to A7); 60 male and 10 female. Each group will consist of 10 subjects of the same sex and 8 subject for DA-8010.
  Part B will comprise a multiple-dose, sequential-group study. Total forty subjects (30 male and 10 female) will be studied in 4 groups (Groups B1 to B4), with each group consisting of 10 subjects of the same sex and 8 subject for DA-8010.
  Arms: Active in Group A1~A7; Active in Group B1~B4
Drug: Placebo — Part A will comprise a single-dose, sequential-group study incorporating a food effect evaluation. Total 70 subjects will be studied in 7 groups (Groups A1 to A7); 60 male and 10 female. Each group will consist of 10 subjects of the same sex and 2 subject for DA-8010.
  Part B will comprise a multiple-dose, sequential-group study. Total forty subjects (30 male and 10 female) will be studied in 4 groups (Groups B1 to B4), with each group consisting of 10 subjects of the same sex and 2 subject for DA-8010.
  Arms: Placebo in Group A1~A7; Placebo in Group B1~B4

SUMMARY:
This study is a Phase I, Randomised, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate Safety, Tolerability and Pharmacokinetics After Single and Multiple Oral Administration of DA-8010 in Healthy Subjects.

DETAILED DESCRIPTION:
This study will be a randomised, double-blind, placebo-controlled, dose-escalation, single and multiple oral dose study conducted in 2 parts.

In Part A, each subject will participate in 1 treatment period only and reside at the Clinical Research Unit (CRU) from Day -1 (the day before dosing) to Day 3 (48 hours postdose), except for Group A4, where each subject will participate in 2 treatment periods separated by a minimum of 13 days to evaluate the effect of food.

In Part B, each subject will participate in 1 treatment period only and reside at the CRU from Day -1 (1 day before dosing) until the morning of Day 9 (48 hours after the final dose on Day 7).

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.0 and 32.0 kg/m2
* Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

* Subjects who do not agree to use a method of acceptable contraception
* Female subjects of child-bearing potential who do not agree to use a highly effective method of birth control
* Consume more than 28 or 21 units of alcohol per week if male or female, respective
* Subjects who have used nicotine-containing products (including cigarettes), within 3 months prior to the first dose administration
* Subjects who have used, or intend to use the product like non-prescribed systemic or topical medication, herbal remedy, vitamin/mineral supplement, within 7 days of the first dose administration
* Systolic blood pressure < 90 mmHg or > 140 mmHg
* Diastolic blood pressure < 50 mmHg or > 90 mmHg
* Pulse rate < 45 bpm or > 100 bpm
* Positive urine drugs of abuse screen at screening or first admission
* Positive alcohol breath test at screening or first admission
* Positive cotinine test at screening or first admission
* Abnormality in the 12-lead ECG at screening, admission or predose on Day 1
* Subjects who are pregnant, breastfeeding, or lactating
* Subjects who are still participating in another clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of any investigational drug in the past 3 months prior to the first dose administration
* Subjects who have a significant history of drug allergy, as determined by the Investigator
* Aspartate aminotransferase and/or Alanine aminotransferase ≥ 1.5 × upper limit of normal (ULN) or total bilirubin > ULN at screening or admission
* Subjects who are carriers of HBsAg or hepatitis C antibody, have serum hepatitis or positive result for the test for HIV antibodies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | during 10 days in Part A
  Safety outcome will be assessed by incidence and severity of several items (adverse events, vital signs, electrocardiography, clinical laboratory evaluations, physical examination).
Safety and Tolerability | during 16 days in Part B
  Safety outcome will be assessed by incidence and severity of several items (adverse events, vital signs, electrocardiography, clinical laboratory evaluations, physical examination).

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | 48 hours
Maximum observed plasma concentration (Cmax) | 48 hours
Time of the maximum observed plasma concentration (tmax) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jisu Song, Study Director — Dong-A ST

IPD SHARING:
Plan to Share IPD: No